CLINICAL TRIAL: NCT03596463
Title: Influence of Multidisciplinary Breast Tutor Board on Physician Clinical Decision
Brief Title: Influence of Multidisciplinary Breast Tumor Board on Physician Decision
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Murat Ferhat Ferhatoglu, Assistant professor, M.D., Okan University
Other Study IDs: OkanU2
Record Dates: First submitted 2018-07-11; First posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer; Breast Neoplasms; Surgery; Oncology
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Patients treated according to suggestions of tumor board
  Interventions: Other: Breast cancer treatment
- Group B: Patients not treated according to suggestions of tumor board
  Interventions: Other: Breast cancer treatment

INTERVENTIONS:
Other: Breast cancer treatment — Multidisciplinary approach for breast cancer treatment is more beneficial for the patients

SUMMARY:
In our study, the treatment plan for the case prior to the breast tumor counseling will be asked to physician and the treatment protocol observed by the primary physician will be observed after the decision of the tumor council.

ELIGIBILITY:
Inclusion Criteria:

Patients having primary breast cancer

Exclusion Criteria:

Patients having recurrent breast cancer -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 120 patients having breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-08-13 (Estimated); Primary Completion 2019-08-13 (Estimated); Study Completion 2019-11-13 (Estimated)

PRIMARY OUTCOMES:
Better survival | 2 years
  Multidisciplinary approach creates better survival

IPD SHARING:
Plan to Share IPD: No